CLINICAL TRIAL: NCT03776045
Title: Effects of Exercise in Prostate Cancer Patients Initiating Androgen Deprivation Therapy: A Randomised Controlled Trial
Brief Title: PROState Cancer Patients Initiating Hormone Therapy: Effect of Exercise on CARDIOvascular Health (PROSCARDIO)
Acronym: PROSCARDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROSCARDIO1992
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen deprivation therapy; Exercise
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Standard of Care; Exercise

STUDY DESIGN:
Intervention Model Description: After baseline measures were collected, participants were randomly allocated (1:1) to standard care or standard care plus exercise using a randomisation sequence created by an independent researcher (nQuery, Statistical Solutions, USA). Treatment allocation was concealed from the research team until after baseline measurements were collected.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts were blind to treatment allocation. It was not possible to blind participants or the intervention facilitator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): This group did not receive any supervised exercise or were not given any specific exercise recommendations during the trial period. However, patients in this group were offered the exercise intervention after completing the study.
- Standard care plus exercise (Experimental): This group received standard care in addition to a 3-month exercise intervention upon initiating androgen deprivation therapy.
  Interventions: Other: Standard care plus exercise

INTERVENTIONS:
Other: Standard care plus exercise — The exercise was supervised by exercise science staff in the exercise science facilities at the University of East Anglia, UK. Participants competed two weekly sessions for 12 weeks upon initiating ADT. Each session lasted ~60 min and included aerobic interval exercise on a cycle ergometer (Monark 824E; Varberg, Sweden) followed by resistance training. In addition to the supervised exercise sessions, patients were advised on how to increase their habitual physical activity levels and were encouraged to engage in 30 minutes of self-directed exercise on three days each week (e.g. brisk walking, cycling, home-based resistance training).
  Arms: Standard care plus exercise

SUMMARY:
This study evaluates whether exercise can reduce treatment-related adverse effects in prostate cancer patients initiating androgen deprivation therapy. Half of recruited participants completed a 3-month exercise intervention, while the other half did not perform any supervised exercise. It was anticipated that exercise would have a positive effect on body composition, cardiorespiratory fitness and quality of life.

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) is routinely used as first-line treatment for locally advanced and metastatic prostate cancer. However, it is associated with many side effects such as increased fat mass and reduced skeletal muscle mass, cardiorespiratory fitness and metabolic health. Ultimately, these negative changes induced by ADT contribute to reduced health-related quality of life (HRQoL). This study evaluates whether 3-months of exercise can mitigate treatment toxicity in prostate cancer patients initiating ADT.

In a parallel groups, prospective, randomised controlled design, participants were randomly allocated to a standard care control group or standard care plus exercise group. The exercise group completed 3-months of combined aerobic and resistance training. The standard care group did not receive any supervised exercise or specific physical activity recommendations. Outcomes were assessed at baseline, 3-month (post-intervention), and 6-month (follow-up) endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 50 to 80 years
* Histologically confirmed stage I-IV prostate cancer
* Scheduled for treatment with a luteinizing hormone-releasing hormone (LHRH) agonist either alone or combined with radiotherapy
* Anticipated to remain on androgen deprivation therapy (ADT) for at least the next 6 months
* Willing and able to give written informed consent.
* Understand written and verbal instructions in English
* World Health Organisation (WHO) performance status 0 to 1

Exclusion Criteria:

* Previously treated with ADT
* Diagnosed or suspected metastatic bone disease
* Absolute contraindications to exercise testing and training as defined by the American College of Sports Medicine (ACSM, 2010)
* Prior myocardial infarction or heart failure
* Chronic obstructive pulmonary disease (COPD)
* Poorly controlled hypertension (≥ 200/110 mmHg)
* Uncontrolled supraventricular tachycardia (≥ 100 bpm)
* Pre-existing severe musculoskeletal, neurological or psychiatric condition that may affect their ability to complete the testing battery or exercise training, as determined by the patient's physician
* Involvement in any other clinical trial or exercise trial

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08-12 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2016-02-03 (Actual)

PRIMARY OUTCOMES:
Whole body fat mass (kg) | Adjusted mean difference between groups at 3-month endpoint
  Whole body fat mass was measured with bioelectrical impedance analysis (BIA) and concurrent bioelectrical impedance vector analysis (BIVA) with a single-frequency, phase-sensitive 50 kilohertz bioelectrical impedance analyzer (BIA-101, RJL/Akern Systems, Florence, Italy). This was chosen as the primary outcome because adiposity has shown a high propensity to increase during the initial phases of androgen deprivation therapy, more so than other measures (Galvao et al. 2011), which highlights the importance of targeting body fat at this stage of treatment.

SECONDARY OUTCOMES:
Whole body fat mass (kg) | Adjusted mean difference between groups at 6-month endpoint
  Whole body fat mass was measured with bioelectrical impedance analysis (BIA) and concurrent bioelectrical impedance vector analysis (BIVA) with a single-frequency, phase-sensitive 50 kilohertz bioelectrical impedance analyzer (BIA-101, RJL/Akern Systems, Florence, Italy). This was chosen as the primary outcome because adiposity has shown a high propensity to increase during the initial phases of androgen deprivation therapy, more so than other measures (Galvao et al. 2011), which highlights the importance of targeting body fat at this stage of treatment.
Whole body fat-free mass (kg) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Whole body fat-free mass was measured with bioelectrical impedance analysis (BIA) and concurrent bioelectrical impedance vector analysis (BIVA) with a single-frequency, phase-sensitive 50 kilohertz bioelectrical impedance analyzer (BIA-101, RJL/Akern Systems, Florence, Italy). This method is highly valid for measuring changes in body composition (Savastano et al. 2010).
Anthropometric measurements (cm) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Waist, hip, mid-upper arm, forearm, mid-thigh and calf circumferences were measured with a non-stretching tape using standard techniques.
Peak oxygen consumption (VO2peak, ml/kg/min) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Determined as the highest oxygen consumption (V̇O2) attained during the cardiopulmonary exercise test
Ventilatory anaerobic threshold (ml/kg/min) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Estimated using the modified V-slope method and confirmed by evaluating ventilatory equivalents and end-tidal pressures. Two analysts independently determined the ventilatory anaerobic threshold, with discrepancies of ≥ 7.5% resolved through discussion and consultation with a third analyst if necessary.
Ventilatory equivalents for O2 (V̇E/V̇O2) and CO2 (V̇E/V̇CO2) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Ratio of minute ventilation to O2 consumption and CO2 output at the ventilatory anaerobic threshold
Oxygen pulse (ml/beat) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Ratio of oxygen consumption to heart rate at peak exercise during the cardiopulmonary exercise test
Oxygen uptake efficiency slope (OUES) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Determined as the linear relationship between oxygen uptake and the logarithmic transformation of minute ventilation during the cardiopulmonary exercise test
Concentration of cholesterol (mmol/L) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Concentrations of total cholesterol, low-density lipoprotein (LDL-C) and high-density lipoprotein (HDL-C) were measured from venous blood.
Concentration of triglycerides (mmol/L) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  The concentration of triglycerides was measured from venous blood.
Concentration of testosterone (nmol/L) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Concentration of total testosterone was measured from venous blood.
Concentration of sex hormone binding globulin (nmol/L) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Concentration of sex hormone binding globulin was measured from venous blood.
QRISK®2-2017 score | Adjusted mean difference between groups at 3-month and 6-month endpoints
  The percent risk of a cardiovascular disease event occurring in the next 10 years was calculated with QRISK®2-2017 Web Calculator (https://qrisk.org/2017). The total score ranges from 0 to 100 %, with higher scores indicating a greater risk of cardiovascular disease.
Gleason score | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Gleason scores were measured from prostate biopsies. A score of 1 to 5 is assigned to the cells that make up the largest area of the tumor and another score of 1 to 5 is assigned to the cells that comprise the next largest area. A total Gleason score is then calculated by adding both of these scores together. Total scores ranged from 2 to 10, with 2 representing the most well-differentiated tumors and 10 the least-differentiated tumors.
Prostate specific antigen (ng/mL) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Concentration of prostate specific antigen was measured from venous blood.
Skinfold thickness (mm) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Skinfold thickness was measured at suprailiac and subscapular sites with a skinfold caliper (Harpenden Skinfold Caliper, Baty International, Sussex, UK).
Hand grip strength (kg) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Hand grip strength was measured with an analogue dynamometer (Takei Scientific Instruments Ltd., Tokyo, Japan).
The Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire (version 4) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Disease-specific health-related quality of life was assessed with the FACT-P 39-item questionnaire (version 4). Each item has a 5-point Likert-like response scale ranging from 0 ("Not at all") to 4 ("Very much"). A total score is calculated as the sum of each score from items 1 to 39, which can range from 0 to 156. Negatively worded items are reverse scored (subtracted from 4) prior to summing so that higher total scores indicate better health-related quality of life.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) scale (version 4) | Adjusted mean difference between groups at 3-month and 6-month endpoints
  Fatigue was assessed with the 13-item FACIT-Fatigue scale (version 4). Each item has a 5-point Likert-like response scale ranging from 0 ("Not at all") to 4 ("Very much"). A total score is calculated as the sum of each score from items 1 to 13, which can range from 0 to 52. Negatively worded items are reverse scored (subtracted from 4) prior to summing so that higher total scores indicate less experience of fatigue.
Godin Leisure-Time Exercise questionnaire | Adjusted mean difference between groups at 3-month and 6-month endpoints
  The Godin Leisure-Time Exercise questionnaire was used to characterise levels of physical activity. The questionnaire contains three items and asks the patient to recall the number of bouts of strenuous, moderate, or mild physical activity that exceed 15 min in duration in which they have engaged in over a typical week. A total score is calculated by multiplying the number of strenuous, moderate, and mild physical activity bouts by weights of 9, 5, and 3, respectively, and summing those values in an overall score that ranges from 0 to 119 in arbitrary units. Higher scores indicate participation in higher levels of physical activity.
Number of recruited participants | Descriptive statistics reported during the two-year recruitment period
  Measured as the number of eligible participants who were eligible and consented to participate in the trial. This will be reported in a Consolidated Standards of Reporting Trials (CONSORT) participant flowchart.
Number of adverse events | Descriptive statistics reported during the 3-month intervention period
  The number of adverse events were recorded to determine the feasibility of the exercise intervention. An adverse event was defined as the occurrence of any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the exercise intervention. The type of adverse events was also noted.
Attrition rate | Descriptive statistics reported during the 3-month intervention period.
  Established as the number of patients in the experimental group who discontinued the exercise intervention
Number of patients who were lost to follow-up | Descriptive statistics reported at 3-month and 6-month endpoints
  In the experimental group, patients lost to follow-up were characterised as those who completed the exercise intervention but did not complete endpoint testing. In the control group, patients lost to follow-up were the number of patients who did not complete endpoint testing.
Average number of exercise sessions completed | Descriptive statistics reported during the 3-month intervention period
  The number of exercise sessions completed by each participant in the intervention group was recorded. These values were than averaged to provide a measure of adherence. The maximum number of exercise sessions that participants could complete was 24, so adherence ranged from 0 to 24 sessions, with higher scores indicating greater adherence.

CONTACTS AND LOCATIONS:
Overall Officials: John Saxton, Saxton, Study Director — Northumbria University; Wilphard Ndjavera, MD, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvao DA, Taaffe DR, Spry N, Joseph D, Newton RU. Acute versus chronic exposure to androgen suppression for prostate cancer: impact on the exercise response. J Urol. 2011 Oct;186(4):1291-7. doi: 10.1016/j.juro.2011.05.055. Epub 2011 Aug 17. PMID 21849187
- [Background] Savastano S, Belfiore A, Di Somma C, Mauriello C, Rossi A, Pizza G, De Rosa A, Prestieri G, Angrisani L, Colao A. Validity of bioelectrical impedance analysis to estimate body composition changes after bariatric surgery in premenopausal morbidly women. Obes Surg. 2010 Mar;20(3):332-9. doi: 10.1007/s11695-009-0006-5. Epub 2009 Oct 28. PMID 19862582

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT03776045/SAP_000.pdf